CLINICAL TRIAL: NCT04916184
Title: Effects of Exercise Training on Diastolic and Systolic Dysfunction in Patients With Chronic Heart Failure
Brief Title: Aerobic Versus Combined Exercise and Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Chaveles, Principal Investigator, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43/28.03.2016
Record Dates: First submitted 2021-05-19; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Diastolic Dysfunction; Heart Failure
Keywords: diastolic dysfunction; exercise training
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise (Active Comparator): effects on diastolic dysfunction in patients with stable chronic heart failure
  Interventions: Other: aerobic exercise; Other: combined exercise
- Combined exercise (Active Comparator): effects on diastolic dysfunction in patients with stable chronic heart failure
  Interventions: Other: aerobic exercise; Other: combined exercise

INTERVENTIONS:
Other: aerobic exercise — exercise training rehabilitation (aerobic exercise with/without strength training)
Other: combined exercise — exercise training rehabilitation (aerobic exercise with/without strength training)

SUMMARY:
Thirty-two stable patients with chronic heart failure participated in an exercise rehabilitation program. They randomly assigned to aerobic exercise (AER) or combined aerobic and strength training (COM). Before and after the program, they underwent a symptom-limited maximal cardiopulmonary exercise testing and serial echocardiography evaluation examining the indices of diastolic dysfunction (DD).

DETAILED DESCRIPTION:
Thirty-two stable patients with chronic heart failure (age: 56 ± 10 years, EF: 32 ± 8%, 88 % men) participated in an exercise rehabilitation program. They randomly assigned to aerobic exercise (AER) or combined aerobic and strength training (COM), based on age and peak oxygen uptake, as stratified randomization criteria. Before and after the program, they underwent a symptom-limited maximal cardiopulmonary exercise testing (CPET) and serial echocardiography assessment to evaluate peak oxygen uptake (VO2peak), peak workload (Wpeak), DD grade, right ventricular systolic pressure (RVSP) and EF.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure

Exclusion Criteria:

* atrial fibrillation COPD

Ages: 36 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of a cardiac rehabilitation program on the diastolic dysfunction in patients with chronic heart failure | three months
  Thirty-two stable patients with chronic heart failure (age: 56 ± 10 years, EF: 32 ± 8%, 88 % men) participated in an exercise rehabilitation program. They randomly assigned to aerobic exercise (AER) or combined aerobic and strength training (COM), based on age and peak oxygen uptake, as stratified randomization criteria. Before and after the program, they underwent a serial echocardiography assessment to evaluate the diastolic dysfunction (DD) grade of the left ventricular.
Evaluation of the impact of a cardiac rehabilitation program on the ejection fraction of the left ventricular in patients with chronic heart failure | three months
  Thirty-two stable patients with chronic heart failure (age: 56 ± 10 years, EF: 32 ± 8%, 88 % men) participated in an exercise rehabilitation program. They randomly assigned to aerobic exercise (AER) or combined aerobic and strength training (COM), based on age and peak oxygen uptake, as stratified randomization criteria. Before and after the program, they underwent a serial echocardiography assessment to evaluate the ejection fraction of the left ventricular.

SECONDARY OUTCOMES:
Evaluation of the impact of a cardiac rehabilitation program on the indices of aerobic exercise capacity of the left ventricular in patients with chronic heart failure | three months
  Thirty-two stable patients with CHF (age: 56 ± 10 years, EF: 32 ± 8%, 88 % men) participated in an exercise rehabilitation program. They randomly assigned to aerobic exercise (AER) or combined aerobic and strength training (COM), based on age and peak oxygen uptake, as stratified randomization criteria. Before and after the program, they underwent a cardiopulmonary exercise test to evaluate VO2peak and Wpeak

CONTACTS AND LOCATIONS:
Locations (1):
- Serafim Nanas, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouchla A, Karatzanos E, Dimopoulos S, Tasoulis A, Agapitou V, Diakos N, Tseliou E, Terrovitis J, Nanas S. The addition of strength training to aerobic interval training: effects on muscle strength and body composition in CHF patients. J Cardiopulm Rehabil Prev. 2011 Jan-Feb;31(1):47-51. doi: 10.1097/HCR.0b013e3181e174d7. PMID 20562711
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Result] Kourek C, Alshamari M, Mitsiou G, Psarra K, Delis D, Linardatou V, Pittaras T, Ntalianis A, Papadopoulos C, Panagopoulou N, Vasileiadis I, Nanas S, Karatzanos E. The acute and long-term effects of a cardiac rehabilitation program on endothelial progenitor cells in chronic heart failure patients: Comparing two different exercise training protocols. Int J Cardiol Heart Vasc. 2020 Dec 24;32:100702. doi: 10.1016/j.ijcha.2020.100702. eCollection 2021 Feb. PMID 33392386